CLINICAL TRIAL: NCT04173117
Title: A Low-energy Meal Replacement Plan for Heart Failure With Preserved Ejection Fraction and Type 2 Diabetes: A Feasibility Study
Brief Title: Feasibility of Low Energy Diet in HFpEF and Type 2 Diabetes
Acronym: ALLEVIATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Major delays attributed to COVID-19 pandemic. Learnings informed design of multi-centre RCT
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0699
Record Dates: First submitted 2019-11-08; First posted 2019-11-21 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-05

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Intervention Model Description: Low energy meal replacement plan for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Low energy meal replacement plan 12 weeks
  Interventions: Dietary Supplement: Low energy meal replacement plan (12 weeks)

INTERVENTIONS:
Dietary Supplement: Low energy meal replacement plan (12 weeks) — Low energy meal replacement plan (12 weeks)

SUMMARY:
Open, Single arm intervention, feasibility study

DETAILED DESCRIPTION:
The aims of the proposed feasibility study are to assess whether a low-energy meal replacement plan (MRP) in patients with HFpEF and T2D:

1. Is acceptable to an older, co-morbid, multi-ethnic population

The secondary objectives are to assess whether a low-energy MRP in patients with HFpEF and T2D may be:

1. associated with improved symptoms
2. likely to lead to favourable cardiovascular reverse remodelling
3. likely to improve functional capacity and quality of life
4. associated with favourable reductions in cardiovascular biomarkers
5. associated with increased physical activity
6. associated with favourable cardiovascular outcomes

All patients will undergo the following assessments at baseline, 12-weeks and 12 months (following MRP):

1. Anthropometry: height, weight, BMI.
2. Haemodynamics: resting heart rate and blood pressure.
3. 6-minute walk test +/- cardiopulmonary exercise test (if able to perform)
4. CMR: contrast enhanced, stress perfusion CMR
5. MLWHFQ
6. WHODAS 2.0 (12-item version)
7. Fasting blood test: full blood count, urea and electrolytes, HbA1c, fasting glucose, BNP, high-sensitivity troponin I, insulin and C-peptide. Plasma (≈35mL) will be stored for future biomarker analysis including metabolomics.
8. Urinalysis for proteinuria and urine protein/creatinine ratio.
9. Body composition; dual-energy X-ray absorptiometry (DEXA) scanning.

12. At the end of the 12-week intervention, participants will be invited to a semi-structured interview to explore qualitative aspects of the study to guide future trial design.

13. At 12 months attendance at cardiac rehabilitation will be reviewed.

The MRP provided by Cambridge Weight Plan® contains ~810 kcal/day (30% protein, 50% carbohydrate, 20% fat). The diet will be stopped, and a maintenance diet re-introduced once 50% excess body weight has been lost, or by 12 weeks, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Established T2D (HbA1c ≥6.5%, duration >3months)
* Obesity (BMI ≥30 or ≥27 kg/m2 if black/south Asian ethnicity)
* Symptoms limiting exercise capacity in normal daily activities (dyspnoea or fatigue) or an established diagnosis of HF
* Diagnosis of HFpEF in accordance with European Society of Cardiology criteria: LV EF >50% with objective evidence of cardiac structural or functional alterations (LV hypertrophy (≥12mm); LV mass index ≥115g/m2 for males and ≥95g/m2 for females; E/e' ≥13 and a mean e' septal and lateral wall <9 cm/s; left atrial volume index >34mL/m2 or reduced global longitudinal strain (>-18%); elevated levels of natriuretic peptides (B-type natriuretic peptide >35pg/mL and/or NT-pro B-type natriuretic peptide >125pg/mL))

Exclusion Criteria:

* Unwilling to undertake MRP (low energy diet)
* HBa1c >10%
* Diabetes duration >12 years
* High-dose insulin requirement: either on full basal-bolus insulin regime or insulin requirement >1U/kg/day
* Have been on insulin treatment >10 years
* Current treatment with anti-obesity drugs
* Diagnosed eating disorder or purging
* Weight loss > 5kg in preceding 3 months (unless related to hospitalisation for HF)
* Absolute contraindications to MRI
* Severe renal impairment eGFR<30ml/min/m2
* Myocardial infarction within preceding 6 months
* History of substance abuse
* Cancer undergoing active treatment
* Unable to consent due to lack of mental capacity
* Pregnancy/considering pregnancy
* People unable to perform activities of daily living independently or unable attend for clinical appointments without a carer/attendant
* Unable to read/understand English sufficiently to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates | 16 weeks
  The number of people approached, recruited and retained

SECONDARY OUTCOMES:
Differences in 6 minute walk test pre- and post intervention | 12 weeks
  Meters walked within 6 minutes
Differences in cardiopulmonary exercise test (peak VO2) pre- and post intervention | 12 weeks
  exercise test on a static bike using minute by minute ventilatory gas analysis
Differences in LV remodelling (indexed LV mass) pre- and post intervention | 12 weeks
  CMR measures of cardiac geometry
Differences in LV function pre- and post intervention | 12 weeks
  CMR measures of cardiac function
Differences in E/A ratio pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in E (cm/s) pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in MV deceleration time (ms) pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in A (cm/s) pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in Septal e' pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in Lateral e' pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in Septal E/e' pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in Lateral E/e' pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in Average E/e' pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in LA volume indexed pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in TR jet velocity (m/s) pre- and post intervention | 12 weeks
  Standard clinical echocardiography
Differences in BMI pre- and post intervention | 12 weeks
  Weighing scales and stadiometer measurement (Kg/m2)
Differences in Bone Mineral Density (g/cm2) pre- and post intervention | 12 weeks
  DEXA scan
Differences in Total Fat mass (g) pre- and post intervention | 12 weeks
  DEXA scan
Differences in Total tissue fat (%) pre- and post intervention | 12 weeks
  DEXA scan
Differences in visceral adipose tissue mass (g) pre- and post intervention | 12 weeks
  DEXA scan
Differences in visceral adipose tissue volume (cm3) pre- and post intervention | 12 weeks
  DEXA scan
Differences in Total lean body mass (g) pre- and post intervention | 12 weeks
  DEXA scan
Difference in World Health Organisation Disability Schedule (WHODAS 2.0) pre- and post intervention | 12 weeks
  Scale 0 - 48 with lower scores indicating better outcome
Difference in Medical Research Council Dyspnoea Scale pre- and post intervention | 12 weeks
  scale 1 - 5 with lower scores indicating better outcome
Difference in Minnesota Living with heart Failure Questionnaire pre- and post intervention | 12 weeks
  Scale 0 - 105 with lower scores indicating better outcome
Differences in Fasting Glucose (mmol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in HbA1c (%) pre- and post intervention | 12 weeks
  Biochemistry
Differences in HbA1c (mmol/mol) pre- and post intervention | 12 weeks
  Biochemistry
Differences in B-type (ng/L) natriuretic peptide pre- and post intervention | 12 weeks
  Biochemistry
Differences in hs-troponin (ng/L) natriuretic peptide pre- and post intervention | 12 weeks
  Biochemistry
Differences in CRP (mg/L), natriuretic peptide pre- and post intervention | 12 weeks
  Biochemistry
Differences in albumin concentration pre- and post intervention | 12 weeks
  Biochemistry
Differences in albumin/creatinine ratio concentration pre- and post intervention | 12 weeks
  Biochemistry
Differences in sodium (mmol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in potassium (mmol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in Urea (mmol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in creatinine (umol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in eGFR (ml/min) pre- and post intervention | 12 weeks
  Biochemistry
Differences in hsTnl(ng/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in hALT (iu/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in ALP (iu/L)pre- and post intervention | 12 weeks
  Biochemistry
Differences in LDL (mmol/L) pre- and post intervention | 12 weeks
  Biochemistry
Differences in kidney function pre- and post intervention | 12 weeks
  Blood analysis for eGFR (ml/min)
Differences in liver function pre- and post intervention | 12 weeks
  Blood analysis for ALP (iu/L)
Differences in the levels of physical activity pre- and post intervention | 12 weeks
  Objectively measured with an accelerometer
Cardiac rehabilitation uptake | 12 months
  The proportion of participants who were offered and attended cardiac rehabilitation following completion of the intervention (%)
The number of participants who experience any Major Adverse Cardiovascular Events (MACE) | 12 weeks
  At any point during the study if a participant experiences a major cardiovascular event this will be recorded and reported to sponsor in line with handling serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Research Centre (Glenfield Hospital), Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No